CLINICAL TRIAL: NCT06350669
Title: App-supported Vestibular Rehabilitation (Randomized Controlled Trial)
Brief Title: App-supported Vestibular Rehabilitation (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Sheba Medical Center (Other Government); Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Yoav Gimon, Principal Investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9576-22-SMC
Record Dates: First submitted 2024-03-23; First posted 2024-04-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Vestibular Disorder; Vestibular Diseases; Vestibular Abnormality
Keywords: Vestibular Rehabilitation; App-Assisted Rehabilitation; Rehabilitation Technologies; Adherence; Compliance
MeSH Terms: conditions — Vestibular Diseases; Patient Compliance

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned to either the intervention group (app-assisted vestibular rehabilitation) or the control group ("standard" vestibular rehabilitation/no app)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-assisted vestibular rehabilitation (Experimental): The patients in this group will undergo standard vestibular rehabilitation treatment with the addition of a phone app that support the treatment program, e.g., providing reminders for exercise, documentation of exercise performance, communication with the therapist, etc.
  Interventions: Device: Vestibular rehabilitation phone application
- Standard vestibular rehabilitation (no app) (No Intervention): The patients in this group will undergo standard vestibular rehabilitation treatment, without using the app.

INTERVENTIONS:
Device: Vestibular rehabilitation phone application — The standard vestibular rehabilitation process, with the support of a phone app throughout the process
  Arms: App-assisted vestibular rehabilitation

SUMMARY:
A randomized controlled trial to assess the efficacy of an app-assisted vestibular rehabilitation in increasing adherence to VR and treatment outcomes

DETAILED DESCRIPTION:
Vestibular Rehabilitation (VR) home exercises, prescribed by physiotherapists, are the main treatment for vestibular dysfunction. However, reports by clinicians indicate that patients do not fully comply with the treatment. Advances in technology and tele-rehabilitation have the potential to facilitate adherence to home exercise, if they are designed to overcome the barriers for practice. We plan to continue and expand our previous feasibility study with the vestibular phone app, in order to examine the effects of an app-assisted VR program on adherence and treatment outcomes. The patients in this study will be randomly assigned to the intervention (app-assisted vestibular rehabilitation) or the control group (standard vestibular rehabilitation, no app).

Tests and measurements for both groups will be done at three time points:

1. Preliminary assessment session (Session 1)- An initial assessment test on the first visit;
2. Secondary assessment session (Session 2)- After 5-6 weeks;
3. Follow-up evaluation session (Session 3)- One month after the secondary assessment session.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over
* Diagnosis with any vestibular disorder that requires a vestibular rehabilitation exercise program
* Physical and cognitive ability to perform vestibular physiotherapy

Exclusion Criteria:

* A physical disability that does not allow for the performance of vestibular physiotherapy
* A diagnosis of a central vestibular disorder caused by structural damage to the brain
* Individuals who are not qualified to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Adherence measures | At the end of Cycle 1 (each cycle is 4-6 weeks)
  Quantitative data on adherence to home exercise will be extracted from users' phone application database (intervention group) or from records in a diary / logs (control group)
Timed up and go (TUG) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  Assesses balance, walking ability and also used as a screening test for the risk of falls by assessing the function of the lower limbs. The individual is required to get up from sitting on a chair, walk 3 meter forward at a normal pace, turn around and return to a sitting position. The examiner times this sequence

SECONDARY OUTCOMES:
Demographics and medical history intake | At the beginning of Cycle 1 (each cycle is 4-6 weeks)
  Characteristics of patients
Vestibular functions- physical examination | At the the beginning of Cycle 1 (each cycle is 4-6 weeks)
  The routine assessment of vestibular functions, with fixation and without fixation. These functions include observation of gait, posture, gaze / detection of spontaneous nystagmus and it's characteristics, Vestibulo-Ocular reflex (VOR), head impulse test, head shaking nystagmus, dix-hallpike test, supine roll test and dynamic visual acuity (DVA)
Oculomotor functions- physical examination | At the the beginning of Cycle 1 (each cycle is 4-6 weeks)
  The routine assessment of oculomotor functions: Saccades, Smooth-Pursuit, Vestibulo-Ocular Reflex cancellation (VORc) test, Convergence, single cover and cover-uncover test
Visual Analogue Scale (VAS) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  Subjective ranking of the severity of symptoms of dizziness and nausea in sitting position, standing and walking
Dizziness Handicap Inventory (DHI) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  The Hebrew version of the Dizziness Handicap Inventory (DHI) questionnaire
Activities-specific Balance Confidence Scale (ABC) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  A questionnaire that measures the patient's level of balance confidence in performing daily activities
Dynamic Gait Index (DGI) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  Assesses patient's ability to maintain balance while walking in the presence of external demands
10-Meters Walk Test (10MWT) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  Estimates walking speed in meters per second of a short distance (10-meter walking distance)
2-Minute Walk Test (2MWT) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  Measures the distance the subject can walk in two minutes, aiming to assess endurance, functional mobility and gait
Dynamic Visual Acuity (DVA) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  Tests visual acuity during head movement, which rely on the behavior of the Vestibulo-ocular reflex (VOR)
Video Head Impulse Test (vHIT) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  A test to evaluate the angular VOR and the function of the superior and inferior vestibular nerves
Suppression Head Impulse Test (SHIMP) | At the beginning of Cycle 1, the end of Cycle 1 and the end of Cycle 2 (each cycle is 4-6 weeks)
  To provide the examiner with complementary information about peripheral vestibular function. This is a sensitive indicator of residual vestibular function as well as the usual VOR (Vestibulo-ocular reflex) gain measure
Exercise difficulty levels and symptoms severity | At the end of Cycle 1 (each cycle is 4-6 weeks)
  Quantitative data exercise difficulty levels and symptoms severity will be extracted from users' phone application database
Cognitive reserve index questionnaire (CRIQ) | By the end of Cycle 1 (each cycle is 4-6 weeks)
  A questionnaire for assessing the degree of cognitive reserve. Cognitive reserve describes the resilience of the brain to damage, and is used to interpret individual differences in susceptibility to cognitive impairment in the presence of brain changes associated with age or disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Gimmon, PhD, Principal Investigator — Sheba Medical Center; University of Haifa
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal Y, Carey JP, Della Santina CC, Schubert MC, Minor LB. Disorders of balance and vestibular function in US adults: data from the National Health and Nutrition Examination Survey, 2001-2004. Arch Intern Med. 2009 May 25;169(10):938-44. doi: 10.1001/archinternmed.2009.66. PMID 19468085
- [Background] Alhabib SF, Saliba I. Video head impulse test: a review of the literature. Eur Arch Otorhinolaryngol. 2017 Mar;274(3):1215-1222. doi: 10.1007/s00405-016-4157-4. Epub 2016 Jun 21. PMID 27328962
- [Background] Brooks D, Davis AM, Naglie G. The feasibility of six-minute and two-minute walk tests in in-patient geriatric rehabilitation. Can J Aging. 2007 Summer;26(2):159-62. doi: 10.3138/cja.26.2.009. PMID 17613447
- [Background] Dannenbaum E, Paquet N, Chilingaryan G, Fung J. Clinical evaluation of dynamic visual acuity in subjects with unilateral vestibular hypofunction. Otol Neurotol. 2009 Apr;30(3):368-72. doi: 10.1097/MAO.0b013e31819bda35. PMID 19318888
- [Background] Des Courtis A, Castrillon R, Haenggeli CA, Delaspre O, Liard P, Guyot JP. Evaluation of subjectivity in the interpretation of videonystagmography. Acta Otolaryngol. 2008 Aug;128(8):892-5. doi: 10.1080/00016480701784957. PMID 18607931
- [Background] Gaikwad, S. B., Mukherjee, T., Shah, P. V., Ambode, O. I., Johnsonb, E. G., & Daher, N. S. (2016). Home exercise program adherence strategies in vestibular rehabilitation: a systematic review. Physical therapy rehabilitation science, 5(2), 53-62
- [Background] Gill-Body KM, Beninato M, Krebs DE. Relationship among balance impairments, functional performance, and disability in people with peripheral vestibular hypofunction. Phys Ther. 2000 Aug;80(8):748-58. PMID 10911413
- [Background] Gopinath B, McMahon CM, Rochtchina E, Mitchell P. Dizziness and vertigo in an older population: the Blue Mountains prospective cross-sectional study. Clin Otolaryngol. 2009 Dec;34(6):552-6. doi: 10.1111/j.1749-4486.2009.02025.x. PMID 20070765
- [Background] Hall CD, Herdman SJ. Reliability of clinical measures used to assess patients with peripheral vestibular disorders. J Neurol Phys Ther. 2006 Jun;30(2):74-81. doi: 10.1097/01.npt.0000282571.55673.ed. PMID 16796772
- [Background] Hall CD, Herdman SJ, Whitney SL, Anson ER, Carender WJ, Hoppes CW, Cass SP, Christy JB, Cohen HS, Fife TD, Furman JM, Shepard NT, Clendaniel RA, Dishman JD, Goebel JA, Meldrum D, Ryan C, Wallace RL, Woodward NJ. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Updated Clinical Practice Guideline From the Academy of Neurologic Physical Therapy of the American Physical Therapy Association. J Neurol Phys Ther. 2022 Apr 1;46(2):118-177. doi: 10.1097/NPT.0000000000000382. PMID 34864777
- [Background] Harrell RG, Schubert MC, Oxborough S, Whitney SL. Vestibular Rehabilitation Telehealth During the SAEA-CoV-2 (COVID-19) Pandemic. Front Neurol. 2022 Jan 20;12:781482. doi: 10.3389/fneur.2021.781482. eCollection 2021. PMID 35126289
- [Background] Kao AC, Nanda A, Williams CS, Tinetti ME. Validation of dizziness as a possible geriatric syndrome. J Am Geriatr Soc. 2001 Jan;49(1):72-5. doi: 10.1046/j.1532-5415.2001.49012.x. PMID 11207845
- [Background] Kaplan DM, Friger M, Racover NK, Peleg A, Kraus M, Puterman M. [The Hebrew dizziness handicap inventory]. Harefuah. 2010 Nov;149(11):697-700, 750, 749. Hebrew. PMID 21250408
- [Background] Legters K, Whitney SL, Porter R, Buczek F. The relationship between the Activities-specific Balance Confidence Scale and the Dynamic Gait Index in peripheral vestibular dysfunction. Physiother Res Int. 2005;10(1):10-22. doi: 10.1002/pri.20. PMID 15991483
- [Background] Lempert T, Bronstein A. Management of common central vestibular disorders. Curr Opin Otolaryngol Head Neck Surg. 2010 Oct;18(5):436-40. doi: 10.1097/MOO.0b013e32833dbd69. PMID 20639762
- [Background] Millar JL, Gimmon Y, Roberts D, Schubert MC. Improvement After Vestibular Rehabilitation Not Explained by Improved Passive VOR Gain. Front Neurol. 2020 Feb 20;11:79. doi: 10.3389/fneur.2020.00079. eCollection 2020. PMID 32153490
- [Background] Mutlu B, Serbetcioglu B. Discussion of the dizziness handicap inventory. J Vestib Res. 2013;23(6):271-7. doi: 10.3233/VES-130488. PMID 24447966
- [Background] Nussbaum R, Kelly C, Quinby E, Mac A, Parmanto B, Dicianno BE. Systematic Review of Mobile Health Applications in Rehabilitation. Arch Phys Med Rehabil. 2019 Jan;100(1):115-127. doi: 10.1016/j.apmr.2018.07.439. Epub 2018 Aug 29. PMID 30171827
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Soto-Varela A, Faraldo-Garcia A, Del-Rio-Valeiras M, Rossi-Izquierdo M, Vaamonde-Sanchez-Andrade I, Gayoso-Diz P, Lirola-Delgado A, Santos-Perez S. Adherence of older people with instability in vestibular rehabilitation programmes: prediction criteria. J Laryngol Otol. 2017 Mar;131(3):232-238. doi: 10.1017/S0022215116009932. Epub 2017 Jan 16. PMID 28088930
- [Background] Tyson S, Connell L. The psychometric properties and clinical utility of measures of walking and mobility in neurological conditions: a systematic review. Clin Rehabil. 2009 Nov;23(11):1018-33. doi: 10.1177/0269215509339004. Epub 2009 Sep 28. PMID 19786420
- [Background] Whitney SL, Hudak MT, Marchetti GF. The activities-specific balance confidence scale and the dizziness handicap inventory: a comparison. J Vestib Res. 1999;9(4):253-9. PMID 10472037
- [Background] Whitney SL, Hudak MT, Marchetti GF. The dynamic gait index relates to self-reported fall history in individuals with vestibular dysfunction. J Vestib Res. 2000;10(2):99-105. PMID 10939685
- [Background] Whitney SL, Marchetti GF, Schade A, Wrisley DM. The sensitivity and specificity of the Timed "Up & Go" and the Dynamic Gait Index for self-reported falls in persons with vestibular disorders. J Vestib Res. 2004;14(5):397-409. PMID 15598995
- [Background] Yardley L, Barker F, Muller I, Turner D, Kirby S, Mullee M, Morris A, Little P. Clinical and cost effectiveness of booklet based vestibular rehabilitation for chronic dizziness in primary care: single blind, parallel group, pragmatic, randomised controlled trial. BMJ. 2012 Jun 6;344:e2237. doi: 10.1136/bmj.e2237. PMID 22674920